CLINICAL TRIAL: NCT00965575
Title: Melatonin and Sleep in Patients With Epilepsy
Brief Title: Pilot Study of Melatonin and Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-1042
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2017-02

CONDITIONS: Epilepsy
Keywords: epilepsy; sleep; seizures; cognition
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Experimental): Subjects will take sustained release melatonin 30 minutes prior to bedtime for four weeks
  Interventions: Drug: Melatonin
- Placebos (Placebo Comparator): Subjects will take a placebo 30 minutes before bedtime for four weeks
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Melatonin — Sustained release formula (Brand: Jigsaw); dosage will be 9mg for all subjects. Taken 30 minutes prior to bedtime for four weeks.
  Other Names: natural supplement
  Arms: Melatonin
Drug: Placebos — Placebo. Taken 30 minutes prior to bedtime for four weeks.
  Other Names: Placebo
  Arms: Placebos

SUMMARY:
The prevalence of epilepsy is 1% in the USA. About 30% of epilepsy patients eventually become refractory to medical treatment. Co morbid conditions are becoming as important as seizure control as these affect overall wellbeing. Sleep related complaints are frequent in them including, frequent arousals, difficulty falling asleep and excessive daytime sleepiness. Polysomnography shows increased arousal index, sleep onset latency, and stage shifts and fragmented REM sleep. Poor sleep efficiency causes daytime fatigue, poor cognition and behavior and can worsen seizure control. Stabilizing sleep may improve seizure control. Melatonin is a naturally occurring hormone in the body involved in the regulation of circadian rhythm and exogenously given, has been shown to decrease sleep onset latency, arousals, and there-by increase sleep efficiency in healthy pediatric patients. Similar data does not exist in the patients with epilepsy. As sleep has important impact on epilepsy and overall functioning, it is important to study effect of melatonin in children with epilepsy.

We propose a randomized double blind placebo controlled trial with a cross-over design. Our hypothesis is that, for patients with epilepsy, administration of melatonin 30 minutes before bedtime for four weeks may:

* Improve the quality of sleep;
* Improve daytime functioning in terms of cognition, behavior and quality of life;
* Decrease epileptic potential. We will use polysomnography, electroencephalogram, psychomotor vigilance task, seizure diary, and questionnaires to assess the effect of melatonin on these domains. This study may help to improve the care of children with epilepsy.

DETAILED DESCRIPTION:
Hypothesis 1: Melatonin treatment improves the quality of sleep in patients with epilepsy.

Various studies evaluating sleep problems in patients with epilepsy using questionnaires have shown that 34-45% patients have sleep related problems [1-3]. Cortesi et al reported that children with seizures had higher sleep difficulties than their siblings and controls[4]. Bedtime difficulties, sleep fragmentation, daytime sleepiness, snoring and parasomnia were reported as sleep problems in this population [2, 4]. Patients with refractory seizures and using multiple antiepileptic drugs(AED) showed worse problems[5]. On polysomnography (PSG) these patients show increased arousal index, increased sleep onset latency, fragmented or reduced REM sleep, increased stage shifts and increased Stage 1 sleep and decreased stage 2 and slow wave sleep. [6-9] Melatonin has been shown to decrease sleep onset latency and increase total sleep time and subjectively improve sleep in healthy individuals.[10-15]. Various studies using fast release and sustained release formulations have suggested improvement in sleep efficiency and decreased arousals as well.[16-18] In a randomized placebo controlled study by Gupta et al[19], Melatonin was shown to subjectively improve sleep in patients with epilepsy. Studies in children with neurodevelopmental delay and autism along with epilepsy have also reported similar findings.[17, 20-23] Rationale: There are significant sleep disturbances in children with epilepsy. Melatonin has been shown to improve sleep in this group of patients. However, all these studies report improvement based on parent report and only one study is placebo-controlled. Our study will assess this in randomized placebo controlled fashion and will provide both subjective and objective improvement in sleep with the primary outcome being improved sleep efficiency on PSG.

Hypothesis 2: Melatonin improves daytime functioning in terms of cognition, behavior and quality of life in the patients with epilepsy.

Poor sleep and epilepsy both have detrimental effect on cognition.[24-27] Melatonin by improving sleep may improve cognitive functioning in these patients.

Some patients with epilepsy have poor behavior and psychiatric function.[28-30] Severity of these problems are related to the worsening of the sleep problems.[2, 4] Melatonin by improving sleep may improve the behavior in these patients.

Epilepsy has negative effect on various aspects of the patients' life including social, behavioral, and academic [31, 32]. Questionnaires have been developed to assess the impact on overall quality of life of the patients [33, 34]. These tools are helpful to quickly and subjectively assess quality of life. Based on these studies, it has been shown that patients with refractory seizures have poor quality of life [33-37] and an improvement is seen if the seizure frequency is decreased.[38-41] There has been only one study reporting quality of life (QOL) after use of melatonin in patients with epilepsy. In this randomized placebo controlled study, significant improvement was seen in the cognitive, anxiety and behavior subscales of the QOLCE after use of melatonin.[42] To date, there are no studies reporting on the effect of melatonin on cognition or behavior in epilepsy patients.

Rationale: Poor behavior, cognition and quality of life have been reported in children with epilepsy and sleep disturbances. By improving the quality of sleep, melatonin will improve all these domains. QOLCE has been validated and used in epilepsy patients and will assess the QOL in these patients. Vigilance is the component of cognition that is most consistently and drastically affected by sleep deprivation. PVT measures "vigilant attention" and has been used widely in adult patients to assess the effect of sleep deprivation on cognition. It has been described as a very sensitive measure to see both acute and chronic effects of sleep deprivation. BASC-PRS has been used to assess behavior in children and is found equally useful in epilepsy patients as child behavior check list (CBCL). It is a sensitive tool to compare changes over shorter time span.

Hypothesis 3: Melatonin treatment decreases epileptic potential. Sleep deprivation has been known to induce seizures and epileptic discharges on EEG[43]. Seizures are also known to occur with change in the depth or rhythmicity of sleep.[43] Patients with epilepsy report sleep deprivation as a significant seizure precipitating factor [44, 45]. In a recent study, Haut et al reported that one hour of additional sleep on the preceding night decreased relative odds of a seizure on the subsequent day to 0.91[46]. In a study Oliveira reported that treatment of obstructive sleep apnea (OSA) decreased interictal epileptiform discharges.[47] The belief that fewer epileptiform discharges represent better seizure control is controversial. But a study suggested that decreasing epileptiform discharges on EEG improves behavior.[48] Studies investigating obstructive sleep apnea in patients with epilepsy have reported improvement in seizure control with treatment of OSA [49-54]. These suggest that stabilizing sleep has a beneficial effect on seizure control.

Many studies that evaluated melatonin in epilepsy patients report overall improvement in seizure control[17, 21], while others report no worsening of seizure control after the use of melatonin[20, 22, 23]. Coppola et al reported inconclusive results with regards to seizure control after melatonin use[55]. However, these studies are not powered to account for variability in seizure occurrence reported with epilepsy patients.

Rationale: There are no randomized controlled studies available to evaluate the effect of melatonin on seizure control in the children with epilepsy. This study will identify the effect of short term use of melatonin compared with placebo and will provide pilot data to evaluate this effect in a larger trial in future.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-11 years (prepubertal based on tanner staging)
* Patients with epilepsy (diagnosis based on ILAE).
* Normal intelligence based on school placement (defined as age appropriate; an IEP due to epilepsy related causes is acceptable as is placement in a higher grade) or IQ>70 (testing done with in 12 months of enrollment)
* No history of significant snoring- loud snoring every night outside of a room with closed door
* Combined score of 30 or more on sleep fragmentation, parasomnia and daytime drowsiness subscales on SBQ.

Exclusion Criteria:

* History of significant snoring- loud snoring every night heard outside of a room with closed door
* Diagnosis of obstructive sleep apnea (OSA) or periodic limb movement disorder on PSG
* Vagus nerve stimulator implanted
* History of a major psychiatric disease (e.g. psychosis, major depression)
* History of autism or pervasive development disorder
* Severe neuro-developmental disabilities, as determined by PI
* Clinically significant systemic organic disease, as determined by PI
* Current use of melatonin or sustained release melatonin
* Prior use of sustained release melatonin
* Current use of any hypnotic medications except for medications used as a rescue treatment for seizures
* Use of psychoactive or stimulant medication for attention deficit disorders
* Subjects with immune disorders, lympho-proliferative disorders, and those taking oral corticosteroids or other immuno-suppressants
* Subject or parent/legal guardian might not be reasonably expected to be compliant with or to complete the study.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2011-06; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sejal Jain, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data at this time.

REFERENCES:
- See also: Sleep Medicine — https://doi.org/10.1016/j.sleep.2015.01.005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment was done from cincinnati children's neurology/epilepsy clinics during the period of June 2011 to Dec 2012.
Pre-assignment Details: Actual enrollment was 11. 10 completed the study
Groups:
- Melatonin First Then Placebo: Subjects will take sustained release melatonin 30 minutes prior to bedtime for four weeks
  Melatonin: Sustained release formula (Brand: Jigsaw); dosage will be 9mg for all subjects.
  Cross over, so subjects who received melatonin in the first phase will receive placebo during the second phase and vice versa.
- Placebo First Then Melatonin: Subjects will take a placebo 30 minutes before bedtime for four weeks
  Melatonin: Sustained release formula (Brand: Jigsaw); dosage will be 9mg for all subjects.
  Cross over, so subjects who received melatonin in the first phase will receive placebo during the second phase and vice versa.
Period: Overall Study
Arm/Group | Melatonin First Then Placebo | Placebo First Then Melatonin
Started | 6 (cross over, total enrolled 11) | 5 (cross over, total enrolled 11)
Completed | 5 | 5
Not Completed | 1 | 0
Not completed — subject unwillingness to swallow study c | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Melatonin First Then Placebo: Subjects will take sustained release melatonin 30 minutes prior to bedtime for four weeks
  Melatonin: Sustained release formula (Brand: Jigsaw); dosage will be 9mg for all subjects.
- Placebo First Then Melatonin: Subjects will take a placebo 30 minutes before bedtime for four weeks
  Melatonin: Sustained release formula (Brand: Jigsaw); dosage will be 9mg for all subjects.
- Total: Total of all reporting groups
Arm/Group | Melatonin First Then Placebo | Placebo First Then Melatonin | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 5 | 11
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Sleep Latency Wakefulness After Sleep Onset (WASO)
Description: Sleep Latency Wakefulness After Sleep Onset (WASO). Calculated as the sum of wake time minutes from sleep onset to the final awakening.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: minutes/night
Groups:
- Melatonin: Melatonin: Sustained release formula (Brand: Jigsaw); dosage will be 9mg for all subjects. Taken 30 minutes prior to bedtime.
- Placebo: Placebo: taken 30 minutes prior to bedtime
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 10 | 10
minutes/night | 42.3 (30.3) | 57.3 (31.6)

2. Secondary Outcome: Seizure Frequency
Description: Seizure frequency was determined by parent/caregiver report on a seizure diary which was filled out after each seizure which is an accepted patient-reported outcome measure. Data is given as number of seizures per month.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: seizures/month
Groups:
- Melatonin: Subjects will take sustained release melatonin 30 minutes prior to bedtime for four weeks
  Melatonin: Sustained release formula (Brand: Jigsaw); dosage will be 9mg for all subjects.
- Placebo: Subjects will take a placebo 30 minutes before bedtime for four weeks
  Melatonin: Sustained release formula (Brand: Jigsaw); dosage will be 9mg for all subjects.
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 10 | 10
seizures/month | 1.4 (3.8) | 2.4 (6.6)

ADVERSE EVENTS:
Arm/Group | Melatonin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Melatonin (N=10) | Placebo (N=10)
Headache (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No